CLINICAL TRIAL: NCT04027036
Title: Clinical Trial to Compare the Immunogenicity of the Inactivated Poliovirus Vaccine (IPV) Administered in Reduced Doses Intramuscularly or Intradermally in Infants at 2 and 4 Months of Age in the Maputo City
Brief Title: Comparison of Immunogenicity of Inactivated Poliovirus Vaccine (IPV) Administered Intramuscularly or Intradermally
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Saúde, Mozambique (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: fIPV-CISPOC
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Polio
Keywords: Vaccine; Polio Virus
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fIPV Intramuscular (Active Comparator): 180 children will receive 0,1 ml of inactivated poliovirus vaccine intramuscularly
  Interventions: Biological: Inactivated poliovirus vaccine in reduced doses
- fIPV Intradermal (Active Comparator): 180 children will receive 0,1ml of inactivated poliovirus vaccine intradermally
  Interventions: Biological: Inactivated poliovirus vaccine in reduced doses

INTERVENTIONS:
Biological: Inactivated poliovirus vaccine in reduced doses — contains the following excipients: 2-phenoxyethanol (2.5 mg), water for injection and diluent solution and phosphate buffer having the following composition: sodium phosphate, sodium chloride, potassium chloride, magnesium sulfate, phenol red and calcium chloride.
  dosage:0,1ml duration: first dose: month 2 of age; second dose: month 4 of age

SUMMARY:
Polio is an acute transmissible disease caused by any of the three polio virus serotypes (types 1, 2 or 3). In Mozambique, polio vaccination is part of the immunization schedule of the expanded vaccination program. The oral vaccine (OPV) is administered at months 0,2,3, and 4 and a single dose of the inactivated poliovirus vaccine (IPV) is given intramuscularly at month 4. In 2016 shortage of IPV supply caused stock-outs and put strain on IPV use for routine immunizations as well as for poliovirus outbreak response. Therefore, assessment of new vaccine regimens using smaller doses of IPV are needed. Administration of fractionated IPV (fIPV), i.e., 1/5 (0.1mL) of the standard dose, intradermally has shown to be safe and to provide an immune response similar to the standard dose of IPV that is currently given intramuscularly. However, intradermal administration of fIPV is technically difficult and many countries are hesitant to adopt fIPV in their routine immunization schedules. Therefore, the investigators need data confirming that the use of the fIPV vaccine intramuscularly is safe and the immune response is not inferior to the use of fIPV intradermally. Study Objective: to compare the immunogenicity of fIPV administered intramuscularly or intradermally in infants at 2 and 4 months of age. Study Hypotheses: the seroconversion rate after administration of one or two doses of fIPV intramuscularly is not inferior to the fIPV intradermally. The priming effect after fIPV administered intramuscularly is not inferior to the fIPV intradermally. Study Methods: This will be a phase II non-inferiority clinical trial. 360 children will be enrolled in two study groups, with prior consent of the parents / guardians. In group I, 180 children will receive 0.1 ml of IPV intramuscularly and in group II 180 children will receive the same dose intradermally. There will not be a group control. The children will be selected at birth at pre-defined health units in Maputo city. The fractional IPV vaccine will be given to children at 2 and 4 months of age during routine vaccinations. In total there will be four study visits, of which the first two are vaccination visits. All visits will be performed at the health units. 1 ml of blood will be collected at each study visit to assess the immune response before and after vaccination. Data will be collected by trained and qualified personnel and in accordance with Good Clinical Practice standards. Adverse events following administration of the vaccine will be monitored and all serious adverse events will be reported to ethics and regulatory committees, and to World Health Organization (WHO). Evaluation of the immune response: Seroconversion rates and priming effect will be evaluated. Serum will be tested for the presence of neutralizing antibodies against poliovirus using standard neutralization assays and immunogenicity will be assessed by titration of anti-polio 2 immunoglobulin G.

ELIGIBILITY:
Inclusion Criteria:

* Children whose parents/guardians consent to their participation;
* Children whose parents/guardians live in the study area and do not intend to depart during the study period.

Exclusion Criteria:

* Children whose parents are under the legal age with exception of 16-years-old parents who are already living in marital status;
* Children whose parents have mental illness;
* Children with immunosuppression.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 382 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion | month 5
  Difference in seroconversion between arms as expressed by proportion of seropositive children on final blood collection.

SECONDARY OUTCOMES:
Priming | month 4+1week
  Difference in priming between arms as expressed by proportion of seropositive children on third blood collection among seronegative children at 2nd bleed

CONTACTS AND LOCATIONS:
Overall Officials: Edna Viegas, MD,PhD, Principal Investigator — INS-CISPOC
Locations (2):
- Mozambique (2):
  - Instituto Nacional de Saúde-Mozambique CISPOC, Maputo
  - INSMozambique, Maputo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Background] Mohammed AJ, AlAwaidy S, Bawikar S, Kurup PJ, Elamir E, Shaban MM, Sharif SM, van der Avoort HG, Pallansch MA, Malankar P, Burton A, Sreevatsava M, Sutter RW. Fractional doses of inactivated poliovirus vaccine in Oman. N Engl J Med. 2010 Jun 24;362(25):2351-9. doi: 10.1056/NEJMoa0909383. PMID 20573923
- [Background] Resik S, Tejeda A, Mach O, Fonseca M, Diaz M, Alemany N, Garcia G, Hung LH, Martinez Y, Sutter R. Immune responses after fractional doses of inactivated poliovirus vaccine using newly developed intradermal jet injectors: a randomized controlled trial in Cuba. Vaccine. 2015 Jan 3;33(2):307-13. doi: 10.1016/j.vaccine.2014.11.025. Epub 2014 Nov 22. PMID 25448109
- [Background] Nelson KS, Janssen JM, Troy SB, Maldonado Y. Intradermal fractional dose inactivated polio vaccine: a review of the literature. Vaccine. 2012 Jan 5;30(2):121-5. doi: 10.1016/j.vaccine.2011.11.018. Epub 2011 Nov 17. PMID 22100886
- [Background] Resik S, Tejeda A, Lago PM, Diaz M, Carmenates A, Sarmiento L, Alemani N, Galindo B, Burton A, Friede M, Landaverde M, Sutter RW. Randomized controlled clinical trial of fractional doses of inactivated poliovirus vaccine administered intradermally by needle-free device in Cuba. J Infect Dis. 2010 May 1;201(9):1344-52. doi: 10.1086/651611. PMID 20350164
- [Background] Cadorna-Carlos J, Vidor E, Bonnet MC. Randomized controlled study of fractional doses of inactivated poliovirus vaccine administered intradermally with a needle in the Philippines. Int J Infect Dis. 2012 Feb;16(2):e110-6. doi: 10.1016/j.ijid.2011.10.002. Epub 2011 Dec 5. PMID 22153001
- [Background] Troy SB, Kouiavskaia D, Siik J, Kochba E, Beydoun H, Mirochnitchenko O, Levin Y, Khardori N, Chumakov K, Maldonado Y. Comparison of the Immunogenicity of Various Booster Doses of Inactivated Polio Vaccine Delivered Intradermally Versus Intramuscularly to HIV-Infected Adults. J Infect Dis. 2015 Jun 15;211(12):1969-76. doi: 10.1093/infdis/jiu841. Epub 2015 Jan 7. PMID 25567841
- [Background] Soonawala D, Verdijk P, Wijmenga-Monsuur AJ, Boog CJ, Koedam P, Visser LG, Rots NY. Intradermal fractional booster dose of inactivated poliomyelitis vaccine with a jet injector in healthy adults. Vaccine. 2013 Aug 12;31(36):3688-94. doi: 10.1016/j.vaccine.2013.05.104. Epub 2013 Jun 13. PMID 23770332
- [Background] Resik S, Tejeda A, Sutter RW, Diaz M, Sarmiento L, Alemani N, Garcia G, Fonseca M, Hung LH, Kahn AL, Burton A, Landaverde JM, Aylward RB. Priming after a fractional dose of inactivated poliovirus vaccine. N Engl J Med. 2013 Jan 31;368(5):416-24. doi: 10.1056/NEJMoa1202541. PMID 23363495
- [Background] Weldon WC, Oberste MS, Pallansch MA. Standardized Methods for Detection of Poliovirus Antibodies. Methods Mol Biol. 2016;1387:145-76. doi: 10.1007/978-1-4939-3292-4_8. PMID 26983734